CLINICAL TRIAL: NCT06606132
Title: Effects of Immersive Virtual Reality on Quality of Life, Stress, Anxiety, Depression and Grip Strength in Fibromyalgia: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Sebastián (Other)
Responsible Party: Principal Investigator, gonzalo arias alvarez, Sr., Universidad San Sebastián
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Fibromyalgia (FM)
Keywords: fibromyalgia; virtual reality; exercise
MeSH Terms: conditions — Fibromyalgia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A single-arm, pre-post-test pilot study was designed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise with virtual reality (Experimental): The virtual reality program consisted of twelve sessions (2 per week for six weeks) of 10 min warm-up plus 15 minutes of exercise with the FitXR game (developed by FITAR LIMITED) on the Oculus Quest 2™ device. The warm-up consisted of moderate-intensity aerobic exercise on a cycle ergometer. The BORG CR-10 perceived exertion scale was used to determine this intensity. Subsequently, they continued with the FitXR game, starting with a 5-minute phase of muscular activation and global movements of their limbs. They performed eye-hand coordination exercises, hitting balls that came to the person at different speeds, and ended with muscle stretching and slow breathing. These exercises presented different difficulty levels and were adjusted to the person's condition. In the same way, as the game developed, it was possible to increase the level and thus increase its complexity.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The virtual reality program consisted of twelve sessions (2 per week for six weeks) of 10 min warm-up plus 15 minutes of exercise with the FitXR game (developed by FITAR LIMITED) on the Oculus Quest 2™ device. The warm-up consisted of moderate-intensity aerobic exercise on a cycle ergometer. The BORG CR-10 perceived exertion scale was used to determine this intensity. Subsequently, they continued with the FitXR game, starting with a 5-minute phase of muscular activation and global movements of their limbs. They performed eye-hand coordination exercises, hitting balls that came to the person at different speeds, and ended with muscle stretching and slow breathing. These exercises presented different difficulty levels and were adjusted to the person's condition. In the same way, as the game developed, it was possible to increase the level and thus increase its complexity.
  Other Names: virtual reality

SUMMARY:
The aim of this pilot study is to determine the effectiveness of an exercise program based on virtual reality on the impact on quality of life, stress, anxiety, depression and grip strength in people with fibromyalgia. The main questions that are intended to be answered are:

Does therapeutic exercise complemented with immersive virtual reality reduce the impact on quality of life, stress, anxiety and depression and grip strength in people with Fibromyalgia?

The investigators will conduct a pilot study with pre- and post-treatment evaluations. This treatment will consist of 12 sessions of aerobic exercise plus exercise with immersive virtual reality.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a chronic rheumatic disorder characterized by widespread musculoskeletal pain, mood problems, and cognitive impairment with a worldwide prevalence ranging from 2 to 4%, affecting mainly women in a 9:1 ratio and with the age of most significant impact between 25 and 50 years. Patients with FM have an impaired quality of life and frequently seek medical attention, which is reflected in significant healthcare costs. It is estimated that the annual number of medical consultations for FM is almost double that of healthy individuals. Although the exact etiology is not yet fully understood, it has been described that people have a genetic predisposition that, together with physical and emotional factors, including the chronicity of a neuromusculoskeletal injury, can trigger it.

The diverse symptomatology of FM makes it challenging to diagnose. Patients often report a feeling of muscle weakness and fatigue, which can diminish their ability to maintain adequate strength for daily tasks. The altered pain perception that characterizes FM can make even simple tasks such as gripping difficult, as pain and discomfort tend to intensify with repetitive or prolonged use of the hand and forearm muscles. Several studies have reported a generalized decrease in muscle strength, noting that this decrease is inversely related to symptom severity. Psychologically, people with FM are characterized by the presence of negative emotions associated with a state of generalized distress. This state of psychological distress can be accompanied by cognitive and emotional disturbances that can considerably affect the quality of life of patients and even the severity of the syndrome. Constant preoccupation with pain management and uncertainty about the future are both associated with additional symptoms, such as difficulty sleeping and fatigue. The above creates a vicious circle in which stress contributes to physical discomfort, and physical discomfort favors stress. In this context, several authors suggest that there may be reduced levels of resilience and effective coping strategies that may generate low self-efficacy and inefficient modulation of nociceptive stimuli, leading to a bidirectional relationship between the presence of pain and psychoemotional symptoms. On the other hand, these psycho-cognitive mechanisms may be influenced by nociplastic and inflammatory alterations, which would contribute to a reciprocal etiopathogenesis between central and peripheral mechanisms, making treatment more difficult.

The 2017 European guideline recommendations for FM propose a multimodal therapeutic approach that can be tailored to the individual patient's characteristics and contributes to reducing symptom severity and improving quality of life, allowing the person to learn to live as well as possible with their disease. This approach starts with non-pharmacological measures such as health education, physical therapy, and psychotherapy, followed by pharmacological measures such as using pain modulators like duloxetine or pregabalin and medications for sleep disorders. Different studies propose that these approaches can be used simultaneously and that other complementary strategies that could improve the patient's therapeutic experience should also be considered.

Virtual reality (VR) systems have proven to be a complementary therapeutic option with beneficial effects for treating various health conditions. One of the modalities that present a relevant multisensory experience corresponds to immersive virtual reality-based exercise (iVRE), which, given the high level of immersion provided by VR, offers a unique experience, becoming a promising tool in the active treatment of FM. Patients enter a controlled virtual environment that can complement or improve conventional treatment. Current evidence describes the efficacy of VR in chronic pain syndromes and central neurological injuries, incorporating relaxation exercises, cognitive therapies, and adapted physical activities. This interaction may improve cognitive function and reduce symptoms of anxiety and depression associated with their health condition.

Although there is a growing body of knowledge associated with favorable experiences in using VR in FM, it is incipient concerning the immersive modality, particularly when coupled with exercise . In fact, a recent systematic review suggests new studies that include the benefits of this intervention on physical capacity, quality of life, and psychoemotional variables in FM. Therefore, this study aims to evaluate the effect of an iVRE program on the impact of FM on quality of life, stress, anxiety, depression, and handgrip strength in people with FM.

A single-arm, pre-post-test pilot study was designed. The study was conducted at the Universidad San Sebastián, Bio Bío, Chile, and originated from a collaborative project of Community Engagement ('Vinculación con el Medio') of the same University. The study sample was recruited by convenience after applying the following criteria: i) Inclusion: Adults over 18 years of age diagnosed with FM. This diagnosis was previously made by a medical professional under the updated FM diagnostic criteria; ii) Exclusion: Women in a state of pregnancy or breastfeeding, oncological pain, uncontrolled metabolic disorder, vertigo or similar condition, or any physical or cognitive impairment that would hinder communication with the investigators and the ability to perform the intervention protocols.

The clinical investigators performed a complete anamnesis and completed a structured clinical form to collect sociodemographic, health, and pharmacological treatment data. The Scientific Ethical Committee of the Universidad San Sebastián approved this study (N° 151-23). It was conducted following the 1964 Declaration of Helsinki and its subsequent modifications. All patients signed an informed consent form prior to participation.

Intervention (iVRE)

The iVRE program consisted of twelve sessions (2 per week for six weeks) of 10 min warm-up plus 15 minutes of exercise with the FitXR game (developed by FITAR LIMITED) on the Oculus Quest 2™ device. The warm-up consisted of moderate-intensity aerobic exercise on a cycle ergometer. The BORG CR-10 perceived exertion scale was used to determine this intensity. Subsequently, they continued with the FitXR game, starting with a 5-minute phase of muscular activation and global movements of their limbs. They performed eye-hand coordination exercises, hitting balls that came to the person at different speeds, and ended with muscle stretching and slow breathing. These exercises presented different difficulty levels and were adjusted to the person's condition. In the same way, as the game developed, it was possible to increase the level and thus increase its complexity.

ELIGIBILITY:
Inclusion Criteria:

-Males and females; over 18 years of age; with a diagnosis of fibromyalgia issued by a medical professional under the ACR criteria (2016)

Exclusion Criteria:

* Subjects were excluded from the study when they presented pregnancy or lactation; oncologic pain; uncontrolled metabolic disorder; vertigo or similar condition or any cognitive impairment that hinders the understanding of the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Impact of Fibromyalgia on Quality of Life | six weeks
  The Impact of Fibromyalgia on Quality of Life was assessed using the FIQ-R instrument. This self-administered test measures difficulty in activities of daily living in the last week, the overall influence of the disease in the last week, and the severity of symptoms in the past week. Total scores range from 0 to 100, with higher scores indicating more severe symptoms and disability

SECONDARY OUTCOMES:
Stress, anxiety and depression | six weeks
  Stress, anxiety, and depression were assessed using the Depression Anxiety Stress Scale-21 (DASS-21). This self-administered dimensional test consists of twenty-one questions to evaluate three categories, specifically stress, anxiety, and depression. It presents four response options for each category, evaluated on a scale from 0 to 3. The score obtained for each category is multiplied by 2, and the result is classified as normal, mild, moderate, severe, and extremely severe
Handgrip strength | six weeks
  The handgrip strength was measured with a Baseline hydraulic dynamometer (Fabrication Enterprises Inc., White Plains, NY). The dominant side was evaluated, and the average of three measurements in kilograms was obtained. The position of each measurement was performed with the subject seated, elbow flexed at 90°, wrist in neutral position, and the subject was instructed to squeeze the instrument as hard as possible.

CONTACTS AND LOCATIONS:
Overall Officials: GONZALO j ARIAS ALVAREZ, Master, Principal Investigator — Universidad San Sebastián
Locations (1):
- Universidad San Sebastián, Concepción, Chile

IPD SHARING:
Plan to Share IPD: Undecided
WE DIDN'T HAVE IT CONSIDERED, BUT WE DON'T RULE OUT IT IN THE FUTURE.